CLINICAL TRIAL: NCT07396376
Title: Protocol ELU42 01 01: Phase I/IIA, Open Label, Single Arm Evaluation of Topical ELU42 (XAV939 in DHA77) for Wagner Grade 1-2 Diabetic Foot Ulcers
Brief Title: Evaluation of ELU42 Topical Spray for the Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eluciderm Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND169928
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Foot Ulcer; Wagner Grade 1 - 2; Chronic Wound; Open Wound
Keywords: Wagner 1 and 2 Ulcer; Chronic Wound; DFU; Open Wound; Wound Healing
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm, open-label treatment with ELU42 topical spray applied to the index diabetic foot ulcer (Experimental)
  Interventions: Drug: ELU42 Topical Spray

INTERVENTIONS:
Drug: ELU42 Topical Spray — Topical spray applied per protocol to the index DFU for up to six weeks. Subjects whose wounds reopen during Healing Confirmation visits may restart a full six-week course (maximum 18 applications). Dose volume and application technique per protocol and pharmacy manual.

SUMMARY:
ELU42 01 01 (SuperHealer42) is a Phase I/IIA open label study sponsored by Eluciderm, Inc. that evaluates the safety and preliminary effectiveness of ELU42, a topical small molecule designed to modulate Wnt signaling, for the treatment of chronic diabetic foot ulcers (DFU). ELU42 combines a tankyrase inhibitor (XAV939) with a novel derivatized hyaluronic acid excipient (DHA77) and is applied as a topical spray to the index ulcer.

Fifteen adults with Wagner grade 1-2 diabetic foot ulcers that have been present for at least 4 weeks and up to 52 weeks will be enrolled across up to four U.S. clinical sites. After a 2 week run in period during which standard of care (SOC) is provided (off loading, dressings, and debridement), subjects will receive ELU42 applied on site by trained study staff or the investigator three times per week (Monday, Wednesday, Friday) for six weeks (up to 18 applications). Subjects will be followed weekly during treatment and for up to 6 weeks after the final dose; additional Healing Confirmation visits are scheduled if the wound closes to evaluate the subjects over a course of a 3 month period.

The study's co-primary objectives are to assess safety (incidence and severity of adverse events and infections) and to measure percent area reduction (PAR) of the index ulcer at Weeks 4 and 6. Efficacy assessments will be performed by the site investigator using direct two axis planimetry and by automated evaluation using the Tissue Analytics platform (surface area, volume, and PAR). Secondary and exploratory assessments include patient reported outcomes (Wound Q and SF 36), frequency of complete wound healing, wound hydration metrics, and pharmacokinetic sampling in a subset of subjects.

Contact information for potential participants and referring clinicians is available at each participating site.

DETAILED DESCRIPTION:
ELU42 is a small molecule Wnt signaling modulator intended to promote wound healing in chronic diabetic foot ulcers. This early-phase, single-arm, open-label study evaluates safety, systemic exposure indicators, and preliminary efficacy. Subjects receive topical ELU42 for up to six weeks. If a healed wound reopens during Healing Confirmation visits, subjects may restart a full six-week treatment course (maximum 18 applications). Safety assessments include CBC, CMP, ECGs, nutritional markers, and reproductive safety monitoring. Efficacy assessments include Percentage Area Reduction (PAR) and complete wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to ≤75 years;
* Diagnosis of type 1 or type 2 diabetes mellitus;
* A1C ≤ 10 (historical within 2 months accepted);
* BMI ≤ 36;
* Index DFU Wagner grade 1-2 with post debridement area ≥1.0 cm2 and ≤8.0 cm2;
* Index DFU present for 4-52 weeks;
* Index ulcer ≥1 cm below malleoli;
* Adequate perfusion per ABI/TcPO2/PVR/TBI or Doppler; plantar ulcers off loaded ≥14 days prior to treatment;
* Ability to consent and attend visits;
* Contraception requirements for females of childbearing potential.

Exclusion Criteria:

* Infected index ulcer or surrounding cellulitis;
* Ischemic ulcers; osteomyelitis or exposed bone;
* Recent systemic antibiotic requirement for active infection (eligibility after resolution and 7 day washout);
* Acute/inactive Charcot preventing off loading; hemoglobin < 10 g/dL (unless Sponsor approves);
* ESRD requiring dialysis;
* Recent/planned vascular procedure on target leg within 30 days;
* Participation in other IP trials within 30 days;
* Active alcohol/substance abuse within 3 months;
* Pregnancy or lactation;
* Other PI judged exclusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Area Reduction (PAR) | week 4 and week 6
  Percent change in wound area from baseline to Week 4 and week 6 measured by validated planimetry.

SECONDARY OUTCOMES:
Complete Wound Closure | week 12
  100% re-epithelialization with no drainage.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Gateway Clinical Trials, O'Fallon, Illinois
  - Independent Clincal Research LLC, Springfield, Illinois
  - Curalta Clinical Trials, Oradell, New Jersey
  - Futuro Clinical Trials, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Summary results will be posted per regulatory requirements.